CLINICAL TRIAL: NCT04713709
Title: A Single-Dose, Bioequivalence Study of FMXIN001 4 mg Microspheres Powder and Narcan® 4 mg/0.1 mL Nasal Spray Under Fasting Conditions
Brief Title: A Single-Dose, Bioequivalence Study of FMXIN001 4 mg Microspheres Powder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nasus Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NP-NAL-004
Record Dates: First submitted 2021-01-11; First posted 2021-01-19 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Opioid Overdose
Keywords: Naloxone; Nasal; Powder
MeSH Terms: conditions — Opiate Overdose | interventions — Naloxone

STUDY DESIGN:
Intervention Model Description: Open-label, single-dose, randomized, two-period, two treatment, two-sequence, crossover, comparative bioavailability study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- FMXIN001 4 mg Naloxone microspheres powder, (Experimental): Naloxone powder nasal spray from Nasus Pharma, Israel
  Interventions: Combination Product: Nasus Pharma FMXIN001; Combination Product: Nasal Naloxone liquid spray
- Narcan® 4 mg/0.1 mL nasal spray (Active Comparator): Naloxone solution nasal spray from Adapt Pharma, Inc., USA
  Interventions: Combination Product: Nasus Pharma FMXIN001; Combination Product: Nasal Naloxone liquid spray

INTERVENTIONS:
Combination Product: Nasus Pharma FMXIN001 — A nasal spray of 4mg Naloxone Hydrochloride powder in a unit dose device
Combination Product: Nasal Naloxone liquid spray — A nasal spray of 4mg/0.1mL Naloxone Hydrochloride solution in a unit dose device
  Other Names: Narcan

SUMMARY:
A Single-Dose, Bioequivalence Study of FMXIN001 4 mg Microspheres Nasal Powder.

DETAILED DESCRIPTION:
A comparison between FMXIN001 4 mg and Narcan® 4 mg/0.1 mL Nasal Spray under Fasting Conditions. A pharmacokinetic study in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking, male and female subjects, 18 years of age or older.
2. BMI ≥18 and ≤30 kg/m2.
3. Females may be of childbearing or non-childbearing potential:

   * Childbearing potential:

     o Physically capable of becoming pregnant
   * Non-childbearing potential:

     * Surgically sterile (i.e., both ovaries removed, uterus removed, or bilateral tubal ligation); and/or
     * Postmenopausal (no menstrual period for at least 12 consecutive months without any other medical cause).
4. Willing to use acceptable, effective methods of contraception.
5. Able to tolerate venipuncture.
6. Be informed of the nature of the study and give written consent prior to any study procedure.

Exclusion Criteria:

* The following exclusion criteria will be assessed at screening (within 28 days prior to the first drug administration):

  1. Known history or presence of clinically significant neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, genitourinary, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
  2. Known or suspected carcinoma.
  3. Known history or presence of hypersensitivity or idiosyncratic reaction to naloxone or any other drug substances with similar activity.
  4. Known history or presence of clinically significant lactose, galactose, or fructose intolerance.
  5. Presence of hepatic or renal dysfunction.
  6. Presence of nostril or septum piercing.
  7. Presence of abnormal nasal anatomy.
  8. Presence of hay fever/seasonal allergy/rhinitis.
  9. Presence of sinusitis.
  10. Presence of nasal symptoms (e.g., blocked and/or runny nose, nasal polyps).
  11. Presence of nasal septum ulcers or perforations, or nasal trauma within 30 days prior to drug administration.
  12. History of nasal surgery.
  13. History of malabsorption within the last year or presence of clinically significant gastrointestinal disease.
  14. History of atopic allergy (e.g., asthma, urticaria, eczematous dermatitis).
  15. Presence of a medical condition requiring regular medication (prescription and/or over-the-counter) with systemic absorption.
  16. History of drug or alcohol addiction requiring treatment.
  17. Any acute illness (e.g., cold/ rhinitis, acute infection) which is considered significant by the Investigator and that has not resolved within 7 days before the first drug administration.
  18. Positive test result for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
  19. Positive test result for urine drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, phencyclidine, and tricyclic antidepressants) or urine cotinine.
  20. Difficulty fasting or consuming standard meals.
  21. Inability to communicate well with the Investigators and staff (i.e., language problem, poor mental development or impaired cerebral function).
  22. Use of tobacco or nicotine-containing products within 6 months prior to drug administration.
  23. Females who:

      * Have discontinued or changed the use of implanted, intrauterine, intravaginal, or injected hormonal contraceptives within 6 months prior to drug administration;
      * Have discontinued or changed the use of oral or patch hormonal contraceptives within 1 month prior to drug administration;
      * Are pregnant (serum hCG consistent with pregnancy); or
      * Are lactating.
  24. Donation or loss of whole blood (including clinical trials):

      * ≥50 mL and <500 mL within 30 days prior to drug administration;
      * ≥500 mL within 56 days prior to drug administration.
  25. Participation in a clinical trial that involved administration of an investigational medicinal product within 30 days prior to drug administration, or recent participation in a clinical investigation that, in the opinion of the Investigator, would jeopardize subject safety or the integrity of the study results.
  26. On a special diet within 30 days prior to drug administration (e.g., liquid, protein, raw food diet).
  27. Have had a tattoo or body piercing within 30 days prior to drug administration.
  28. Have clinically significant findings in vital signs measurements.
  29. Systolic blood pressure increase or decrease in value by more than 20 mmHg and/or diastolic blood pressure decrease in value by more than 10 mmHg from supine or sitting to standing position.
  30. Have clinically significant findings in a 12-lead ECG.
  31. Have clinically significant abnormal laboratory values.
  32. Have significant diseases.
  33. Have clinically significant findings from a physical examination.
  34. Use of any enzyme-modifying drugs known to induce/inhibit hepatic drug metabolism or alter gastrointestinal pH/movement (e.g., omeprazole, ranitidine) within 30 days prior to drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Unconjugated naloxone in plasma - Cmax | 0 to 8 hours post dose
  Pharmacokinetic Parameters
Unconjugated naloxone in plasma - AUC | 0 to 8 hours post dose
  Pharmacokinetic Parameters
Unconjugated naloxone in plasma - Tmax | 0 to 8 hours post dose
  Pharmacokinetic Parameters
Unconjugated naloxone in plasma - K el | 0 to 8 hours post dose
  Pharmacokinetic Parameters
Unconjugated naloxone in plasma- T half | 0 to 8 hours post dose
  Pharmacokinetic Parameters

SECONDARY OUTCOMES:
Blood pressure | pre-dose
  Safety Monitoring: Vital signs
Pulse | pre-dose
  Safety Monitoring: Vital signs
Blood pressure | 1 hour post dose
  Safety Monitoring: Vital signs
Pulse | 1 hour post dose
  Safety Monitoring: Vital signs
Blood pressure | 2 hour post dose
  Safety Monitoring: Vital signs
Pulse | 2 hour post dose
  Safety Monitoring: Vital signs
Blood pressure | 4 hour post dose
  Safety Monitoring: Vital signs
Pulse | 4 hour post dose
  Safety Monitoring: Vital signs
Blood pressure | 12 hour post dose
  Safety Monitoring: Vital signs
Pulse | 12 hour post dose
  Safety Monitoring: Vital signs
12-Lead ECG | pre-dose
  Safety Monitoring
12-Lead ECG | 0.5 hours
  Safety Monitoring
12-Lead ECG | 2 hours
  Safety Monitoring
12-Lead ECG | 12 hours
  Safety Monitoring
4-item NHANES Pocket Smell Test | pre-dose
  Safety Monitoring
4-item NHANES Pocket Smell Test | 24 hours post dose
  Safety Monitoring
Nasal examination | pre-dose
  Safety Monitoring
Nasal examination | 1 hour
  Safety Monitoring
Nasal examination | 23 hour
  Safety Monitoring
Adverse events | 0 to 24 hour post dose
  Safety Monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Janice Faulknor, MD, CCFP, Principal Investigator — Pharma Medica Research Inc. Canada
Locations (1):
- Pharma Medica Research Inc, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lapidot T, Bouhajib M, Faulknor J, Khan S, Krayz GT, Abrutzky C, Megiddo D. A Novel Faster-Acting, Dry Powder-Based, Naloxone Intranasal Formulation for Opioid Overdose. Pharm Res. 2022 May;39(5):963-975. doi: 10.1007/s11095-022-03247-5. Epub 2022 Apr 6. PMID 35386013
- See also: Lapidot, Tair, et al. "A Novel Faster-Acting, Dry Powder-Based, Naloxone Intranasal Formulation for Opioid Overdose." Pharmaceutical Research (2022): 1-13. — https://link.springer.com/article/10.1007/s11095-022-03247-5